CLINICAL TRIAL: NCT00492427
Title: Correction and Maintenance Study of Subcutaneous Injections of R744 to Predialysis Patients ( Phase III, Comparative Study in Comparison With Epoetin Beta)
Brief Title: Clinical Study of R744 to Predialysis Patients( Phase III, Comparative Study in Comparison With Epoetin Beta)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chugai Pharmaceutical (Industry)
Responsible Party: Takanori Baba, Chugai Pharmaceutical
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JH20565
Record Dates: First submitted 2007-06-26; First posted 2007-06-27 (Estimated); Last update posted 2009-01-08 (Estimated); Status verified 2009-01

CONDITIONS: Predialysis Patients
MeSH Terms: interventions — epoetin beta

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Active Comparator)
  Interventions: Drug: Epoetin beta
- 1 (Experimental)
  Interventions: Drug: R744

INTERVENTIONS:
Drug: R744 — 25μg(s.c.)/2weeks until Hb concentration reaches to 10g/dL or above and the increasing amount of Hb concentration reaches to 1.0g/dL or above, then 25~250μg(s.c.)/4week for 24~26weeks in total.
  Arms: 1
Drug: Epoetin beta — 6000IU(s.c.)/week until Hb concentration reaches to 10.0g/dL or above and the increasing amount of Hb concentration reaches to 1.0g/dL or above,then 3000k~12000IU(s.c.)/2week for 24~26weeks in total.
  Arms: 2

SUMMARY:
This study used as the comparative drug (epoetin beta) will assess the efficacy and safety of subcutaneous R744 in renal anemia patients on Predialysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose serum creatinine level has been ≥ 2.0 mg/dL or creatinine clearance has been ≤ 30 mL /min at any one time point within 12 weeks before registration
* Patients aged ≥ 20 years at the time of obtaining consent
* Patients who have been not receiving a rHuEPO preparation at least 16 weeks before registration
* Patients whose value of Hb concentrations determined the nearest week before registration has been < 10.0 g/dL
* Patients whose transferrin saturation has been ≥ 20 % or ferritin has been ≥ 100ng/mL at any time point within 8 weeks before registration

Exclusion Criteria:

* Patients with hardly controllable hypertension (patients whose diastolic blood pressure has been ≥ 100 mmHg on more than 1/3 of the determining occasions within 12 weeks before registration)
* Patients with congestive cardiac failure (≥ Class III in NYHA cardiac function classification)
* Female patients who are pregnant, lactating, possibly pregnant or not willing to take a contraceptive measure in the period from the day of starting the treatment with the study drug to 90 days after the day of the last dose of the study drug
* Patients with complication of myocardial infarction, pulmonary infarction or cerebral infarction (excluding asymptomatic cerebral infarction)
* Patients confirmed to have serious allergy or serious drug allergy (shock, anaphylactoid symptom)
* Patients hypersensitive to a rHuEPO preparation
* Patients with malignant tumor (including hemic malignant tumor), severe infection, systemic hemic disease (osteomyelodysplasia syndrome, hemoglobinopathy, etc.), hemolytic anemia or apparent hemorrhagic lesion such as digestive tract hemorrhage
* Patients who have received an anabolic hormone preparation, testosterone enanthate or mepitiostane within 12 weeks before registration
* Patients who have received another investigational drug within 12 weeks before registration
* Patients who have received R744 before registration
* Patients whose AST(GOT) value ≥ 100 IU/L or ALT(GPT) value ≥ 100 IU/L before registration
* Patients who have received erythrocyte transfusion within 16 weeks before registration
* Patients for whom a surgical operation accompanied by marked bleeding is planned during the study period
* In addition, patients who are judged as ineligible to participate in this study by the investigator or subinvestigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2007-06; Primary Completion 2008-01 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Rate of patients who maintain mean Hb concentration in the range of ≥ 10.0g/dL and ≤ 12.0g/dL | 26 weeks

SECONDARY OUTCOMES:
Mean Hb concentration for term of evaluation | 26 weeks
The ratio of patients whose Hb concentration reach ≥ 10.0g/dL and increasing amount of Hb concentration reach ≥ 1.0g/dL | 26 weeks
Time required for reaching Hb concentration of ≥ 10.0 g/dL and reaching increasing amount of Hb concentration of ≥ 1.0g/dL | 26 weeks
Slope of regression line of Hb concentration per week | 26 weeks
Variation of QOL | 26 weeks
Adverse events | 26 weeks
Laboratory measurements | 26 weeks
Vital signs, standard 12-lead ECG | 26 weeks
Anti-R744 antibody titer | 26 weeks
Anti-Epoetin beta antibody titer | 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Takanori Baba, Study Chair — Chugai Pharmaceutical,Clinical Research Department 2
Locations (6):
- Japan (6):
  - Chugoku/Shikoku region, Chugoku/Shikoku
  - Chubu region, Chūbu
  - Hokkaido/Tohoku region, Hokkaido/Tohoku
  - Kanto/Koshinetsu region, Kanto/Koshinetsu
  - Kinki/Hokuriku region, Kinki/Hokuriku
  - Kyusyu region, Kyusyu

REFERENCES:
- [Derived] Chung EY, Palmer SC, Saglimbene VM, Craig JC, Tonelli M, Strippoli GF. Erythropoiesis-stimulating agents for anaemia in adults with chronic kidney disease: a network meta-analysis. Cochrane Database Syst Rev. 2023 Feb 13;2(2):CD010590. doi: 10.1002/14651858.CD010590.pub3. PMID 36791280